CLINICAL TRIAL: NCT04188730
Title: A Study to Evaluate the Relative Bioavailability of a Test Formulation of Lofexidine Granules for Reconstitution and the Effect of Food on the Bioavailability of the Test Formulation in Healthy Adult Subjects
Brief Title: A Study Evaluating the Relative Bioavailability of Lofexidine Granules for Reconstitution Compared to LUCEMYRA (Lofexidine) Tablets and the Effect of Food on the Bioavailability of the Lofexidine Granules for Reconstitution
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: USWM, LLC (dba US WorldMeds) (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: USWM-LX2-1001; R01DA047690 (NIH)
Record Dates: First submitted 2019-11-25; First posted 2019-12-06 (Actual); Results first posted 2022-06-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-05

CONDITIONS: Normal Healthy Volunteers
MeSH Terms: interventions — lofexidine; Tablets

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lofexidine (granules for reconstitution), fasted (Experimental): Participants will be administered lofexidine granules for reconstitution following an overnight fast of at least 10 hours.
  Interventions: Drug: Lofexidine (granules for reconstitution)
- LUCEMYRA (lofexidine) tablets, fasted (Active Comparator): Participants will first be administered LUCEMYRA (lofexidine) tablets following an overnight fast of at least 10 hours
  Interventions: Drug: LUCEMYRA (lofexidine) tablets
- Lofexidine (granules for reconstitution), fed (Experimental): Participants will first be administered lofexidine granules for reconstitution, 30 minutes following a standardized breakfast preceded by an overnight fast of at least 10 hours.
  Interventions: Drug: Lofexidine (granules for reconstitution)

INTERVENTIONS:
Drug: Lofexidine (granules for reconstitution) — All subjects will be administered one 0.36 mg dose of lofexidine granules for reconstitution.
  Arms: Lofexidine (granules for reconstitution), fasted; Lofexidine (granules for reconstitution), fed
Drug: LUCEMYRA (lofexidine) tablets — All subjects will be administered one 0.36 mg dose of LUCEMYRA (lofexidine) tablets.
  Arms: LUCEMYRA (lofexidine) tablets, fasted

SUMMARY:
The purpose of this open-label, single-dose, randomized, three-treatment, three-period, four-sequence, crossover study is to evaluate the relative bioavailability of a test formulation of lofexidine granules for reconstitution (oral) and LUCEMYRA tablets under fasted conditions and to evaluate the effect of food on the relative bioavailability of lofexidine granules for reconstitution (oral) when administered under fed compared to fasted conditions.

ELIGIBILITY:
Inclusion Criteria

1. Males and females, 18-50 years of age, inclusive, with a Body Mass Index (BMI) of 20.0-35.0 kg/m², inclusive.
2. Female subjects must meet at least one of the following criterion:

   * Agree to abstain from sexual intercourse from screening and throughout the duration of the study.
   * Have used and agree to continue to use a reliable method of contraception (e.g., condom with spermicide, IUD, hormonal contraceptives) for at least 30 days before initial dosing and throughout the duration of the study.
   * Surgically sterile (bilateral oophorectomy or hysterectomy, bilateral tubal ligation or Essure® device placement at least 3 months prior to initial dosing).
   * At least 1 year postmenopausal and have a documented FSH level ≥ 40 mIU/mL at screening.
3. Good health as determined by lack of clinically significant abnormalities in health assessments performed at screening.
4. Signed and dated informed consent form, which meets all criteria of current FDA regulations.

Exclusion Criteria

1. Females who are pregnant, lactating, or likely to become pregnant during the study.
2. History of allergy or sensitivity to lofexidine or any component of the study drug or history of any drug hypersensitivity or intolerance which, in the opinion of the Investigator, would compromise the safety of the subject or the study.
3. Significant history or current evidence of chronic infectious disease, system disorders, or organ dysfunction, especially cardiovascular disorders (e.g., severe coronary insufficiency, recent myocardial infarction [within 1 year before initial dosing], cerebrovascular disease), respiratory disorders, congenital long QT syndrome, diabetes, hepatic or renal disorders (e.g., chronic renal failure).
4. Pulse < 50 bpm or symptomatic bradycardia, as determined by the Investigator.
5. Clinically significant history of hypotension, as determined by the Investigator, or has a sitting/supine systolic blood pressure < 90 mmHg and/or diastolic blood pressure < 60 mmHg, or hypertension, as determined by the Investigator, or has sitting/supine systolic blood pressure > 190 mmHg and/or diastolic > 95 mmHg; determined at screening.
6. Experiences reduction of systolic blood pressure of at least 20 mmHg or diastolic blood pressure of at least 10 mmHg within 3 minutes of standing from a resting (sitting or supine) position; determined at screening.
7. 12-lead ECG, conducted in triplicate, considered by the Investigator to be clinically significant (e.g., second or third degree heart block, uncontrolled arrhythmia) or has a QTcF (Fridericia's correction) interval > 440 msec in 2 of the 3 ECGs performed; determined at screening.
8. Clinically significant history or presence of any gastrointestinal disease or history of malabsorption within the last year, as determined by the Investigator.
9. History of any psychiatric disorders occurring within the last two years that required the subject to be hospitalized or treated with medication.
10. Subject has history of suicidality based on responses provided on the Columbia-Suicide Severity Rating Scale (C-SSRS), or is at risk for self-harm or harm to others based on clinical interview, at the discretion of the Investigator.
11. Ingestion of grapefruit-containing food or beverages (e.g., Fresca®) within 7 days before dosing.
12. Drug or alcohol addiction requiring treatment in the 12 months before initial dosing.
13. History of excessive alcohol consumption (on average more than 14 units of alcohol/week) during the past 12 months.
14. Positive test results for HIV, Hepatitis B surface antigen, or Hepatitis C antibody.
15. Positive test results for drugs of abuse (benzodiazepines, cocaine, cannabinoids/THC, opiates and at screening only: amphetamines, barbiturates, methadone and phencyclidine).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim New, Study Director — USWM, LLC (dba US WorldMeds)
Locations (1):
- Novum Pharmaceutical Research Services, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Treatment B, Treatment A, Treatment C: Treatment B = LUCEMYRA tablets - fasted conditions Treatment A = Lofexidine granules - fasted conditions Treatment C = Lofexidine granules - fed conditions Participants in Sequence 1 were first administered (Period 1) one 0.36 mg dose of LUCEMYRA (lofexidine) tablets following an overnight fast of at least 10 hours (Treatment B). Following a 7 day interval between doses, participants were administer (Period 2) one 0.36 mg dose of lofexidine granules for reconstitution following an overnight fast of at least 10 hours (Treatment A). Following a 7 day interval between doses, participants were administered (Period 3) one 0.36 mg dose of lofexidine granules for reconstitution, 30 minutes following a standardized high-fat, high-calorie breakfast preceded by an overnight fast of at least 10 hours (Treatment C).
- Sequence 2: Treatment B, Treatment C, Treatment A: Treatment B = LUCEMYRA tablets - fasted conditions Treatment C = Lofexidine granules - fed conditions Treatment A = Lofexidine granules - fasted conditions Participants in Sequence 2 were first administered (Period 1) one 0.36 mg dose of LUCEMYRA (lofexidine) tablets following an overnight fast of at least 10 hours (Treatment B). Following a 7 day interval between doses, participants were administer (Period 2) one 0.36 mg dose of lofexidine granules for reconstitution, 30 minutes following a standardized high-fat, high-calorie breakfast preceded by an overnight fast of at least 10 hours (Treatment C). Following a 7 day interval between doses, participants were administered (Period 3) one 0.36 mg dose of lofexidine granules for reconstitution following an overnight fast of at least 10 hours (Treatment A).
- Sequence 3: Treatment A, Treatment C, Treatment B: Treatment A = Lofexidine granules - fasted conditions Treatment C = Lofexidine granules - fed conditions Treatment B = LUCEMYRA tablets - fasted conditions Participants in Sequence 3 were first administered (Period 1) one 0.36 mg dose of lofexidine granules for reconstitution following an overnight fast of at least 10 hours (Treatment A). Following a 7 day interval between doses, participants were administer (Period 2) one 0.36 mg dose of lofexidine granules for reconstitution, 30 minutes following a standardized high-fat, high-calorie breakfast preceded by an overnight fast of at least 10 hours (Treatment C). Following a 7 day interval between doses, participants were administered (Period 3) one 0.36 mg dose of LUCEMYRA (lofexidine) tablets following an overnight fast of at least 10 hours (Treatment B).
- Sequence 4: Treatment C, Treatment A, Treatment B: Treatment C = Lofexidine granules - fed conditions Treatment A = Lofexidine granules - fasted conditions Treatment B = LUCEMYRA tablets - fasted conditions
  Participants in Sequence 4 were first administered (Period 1) one 0.36 mg dose of lofexidine granules for reconstitution, 30 minutes following a standardized high-fat, high-calorie breakfast preceded by an overnight fast of at least 10 hours (Treatment C). Following a 7 day interval between doses, participants were administer (Period 2) one 0.36 mg dose of lofexidine granules for reconstitution following an overnight fast of at least 10 hours (Treatment A). Following a 7 day interval between doses, participants were administered (Period 3) one 0.36 mg dose of LUCEMYRA (lofexidine) tablets following an overnight fast of at least 10 hours (Treatment B).
Period: Overall Study
Arm/Group | Sequence 1: Treatment B, Treatment A, Treatment C | Sequence 2: Treatment B, Treatment C, Treatment A | Sequence 3: Treatment A, Treatment C, Treatment B | Sequence 4: Treatment C, Treatment A, Treatment B
Started | 4 | 4 | 4 | 4
Period 1 | 4 | 4 | 4 | 4
Period 2 | 3 | 4 | 4 | 4
Period 3 | 3 | 4 | 4 | 4
Completed | 3 | 4 | 4 | 4
Not Completed | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This is a crossover study with an enrollment of sixteen (16) healthy adult subjects. Each subject was eligible to participate in all 3 treatment group (Treatment A, Treatment B, Treatment C).
Groups:
- All Study Participants: 16 individuals were enrolled in this crossover study. Each subject was eligible to participate in all 3 Treatment Groups (Treatment A, Treatment B, Treatment C).
Arm/Group | All Study Participants
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.5 (3.2)
Height [Mean (Standard Deviation); unit: cm] | 175.1 (8.4)
Weight [Mean (Standard Deviation); unit: kg] | 88.0 (14.6)
Tobacco Users [Number; unit: Count of participants]
  Yes | 0
  No | 16

OUTCOME MEASURES:

1. Primary Outcome: Mean Maximum Plasma Concentration (Cmax)
Description: The peak exposure plasma concentrations (Cmax) of lofexidine were observed and measured.
Time Frame: Mean from Day 1 through Day 3 for Periods I, II, III.
Population: Only sufficient data for 15 of the 16 participants to be analyzed for Pharmacokinetic data due to one participant dropping out after Sequence 1 of the study.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Treatment A: Lofexidine Granules - Fasted Conditions: Participants will be administered lofexidine granules for reconstitution following an overnight fast of at least 10 hours.
  Lofexidine (granules for reconstitution): All subjects will be administered one 0.36 mg dose of lofexidine granules for reconstitution.
- Treatment B: LUCEMYRA Tablets - Fasted Conditions: Participants will first be administered LUCEMYRA (lofexidine) tablets following an overnight fast of at least 10 hours
  LUCEMYRA (lofexidine) tablets: All subjects will be administered one 0.36 mg dose of LUCEMYRA (lofexidine) tablets.
- Treatment C: Lofexidine Granules - Fed Conditions: Participants will first be administered lofexidine granules for reconstitution, 30 minutes following a standardized high-fat, high-calorie breakfast preceded by an overnight fast of at least 10 hours.
  Lofexidine (granules for reconstitution): All subjects will be administered one 0.36 mg dose of lofexidine granules for reconstitution.
Arm/Group | Treatment A: Lofexidine Granules - Fasted Conditions | Treatment B: LUCEMYRA Tablets - Fasted Conditions | Treatment C: Lofexidine Granules - Fed Conditions
Number analyzed (Participants) | 15 | 15 | 15
ng/mL | 0.6984 (0.1661) | 0.7275 (0.1657) | 0.6977 (0.1656)

2. Primary Outcome: Time to Maximum Plasma Concentration (Tmax)
Description: Time to peak plasma concentration (h) collection time at which Cmax is first observed.
Time Frame: Day 1 through Day 3 for Periods I, II, III.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment A: Lofexidine Granules - Fasted Conditions | Treatment B: LUCEMYRA Tablets - Fasted Conditions | Treatment C: Lofexidine Granules - Fed Conditions
Number analyzed (Participants) | 15 | 15 | 15
hours | 4.2678 (1.3894) | 4.3367 (1.2364) | 4.5344 (1.6435)

3. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of Last Measurable Concentration (AUC0-t)
Description: Areas under the plasma concentration-time curve from time zero to the time of last measurable concentration (AUC0-t)
Time Frame: Day 1 through Day 3 for Periods I, II, III.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- Treatment A: Lofexidine Granules - Fasted Conditions: Participants were administer one-0.36 mg dose of Lofexidine granules for reconstitution following an overnight fast of at least 10 hours.
- Treatment B: LUCEMYRA Tablets - Fasted Conditions: Participants will first be administered one-0.36 mg dose of LUCEMYRA (lofexidine) tablets following an overnight fast of at least 10 hours.
- Treatment C: Lofexidine Granules - Fed Conditions: Participants will first be administered one-0.36 mg dose of lofexidine granules for reconstitution, 30 minutes following a standardized high-fat, high-calorie breakfast preceded by an overnight fast of at least 10 hours.
Arm/Group | Treatment A: Lofexidine Granules - Fasted Conditions | Treatment B: LUCEMYRA Tablets - Fasted Conditions | Treatment C: Lofexidine Granules - Fed Conditions
Number analyzed (Participants) | 15 | 15 | 15
h*ng/mL | 12.1333 (4.965) | 12.2450 (4.142) | 12.4540 (4.517)

4. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Time Infinity (AUC0-∞)
Time Frame: Mean from Day 1 through Day 3 for Periods I, II, III.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h·ng/mL
Arm/Group | Treatment A: Lofexidine Granules - Fasted Conditions | Treatment B: LUCEMYRA Tablets - Fasted Conditions | Treatment C: Lofexidine Granules - Fed Conditions
Number analyzed (Participants) | 15 | 15 | 15
h·ng/mL | 14.9643 (6.063) | 14.7229 (4.411) | 14.9004 (5.021)

5. Primary Outcome: First-order Terminal Rate Constant (λz)
Time Frame: Mean from Day 1 through Day 3 for Periods I, II, III.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h^-1
Arm/Group | Treatment A: Lofexidine Granules - Fasted Conditions | Treatment B: LUCEMYRA Tablets - Fasted Conditions | Treatment C: Lofexidine Granules - Fed Conditions
Number analyzed (Participants) | 15 | 15 | 15
h^-1 | 0.0549 (0.0150) | 0.0524 (0.0071) | 0.0524 (0.0075)

6. Primary Outcome: First-order Terminal Half-life (T½)
Time Frame: Mean from Day 1 through Day 3 for Periods I, II, III.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment A: Lofexidine Granules - Fasted Conditions | Treatment B: LUCEMYRA Tablets - Fasted Conditions | Treatment C: Lofexidine Granules - Fed Conditions
Number analyzed (Participants) | 15 | 15 | 15
hours | 13.5577 (3.901) | 13.4681 (1.881) | 13.5008 (2.068)

7. Secondary Outcome: Occurrence of Adverse Events (AEs)
Description: Number of Subjects dosed for each Treatment groups: Treatment A = 15 subjects dosed; Treatment B = 16 subjects dosed; Treatment C = 15 subjects dosed
Time Frame: Total from occurrences assessed daily after each dosing for Periods 1-3, as well as end of study (22 days)
Measure: Number; unit: adverse events
Arm/Group | Treatment A: Lofexidine Granules - Fasted Conditions | Treatment B: LUCEMYRA Tablets - Fasted Conditions | Treatment C: Lofexidine Granules - Fed Conditions
Number analyzed (Participants) | 15 | 16 | 15
adverse events | 3 | 13 | 14

ADVERSE EVENTS:
Time Frame: Daily after each dosing for Periods 1-3, as well as End of Study Day 3 Period 3 (22 days)
Description: Number of Subjects dosed for each Treatment groups: Treatment A = 15 subjects dosed; Treatment B = 16 subjects dosed; Treatment C = 15 subjects dosed
Arm/Group | Treatment A: Lofexidine Granules - Fasted Conditions | Treatment B: LUCEMYRA Tablets - Fasted Conditions | Treatment C: Lofexidine Granules - Fed Conditions
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 3/15 | 8/16 | 7/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: Lofexidine Granules - Fasted Conditions (N=15) | Treatment B: LUCEMYRA Tablets - Fasted Conditions (N=16) | Treatment C: Lofexidine Granules - Fed Conditions (N=15)
Blood pressure decreased (Investigations) | 2 | 4 | 4
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 4 | 3
Dizziness (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2
Pain (General disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/30/NCT04188730/Prot_001.pdf
  • Statistical Analysis Plan (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/30/NCT04188730/SAP_002.pdf
  • Informed Consent Form (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/30/NCT04188730/ICF_000.pdf